CLINICAL TRIAL: NCT01694771
Title: A Randomised, Double Blind, Parallel Group Study to Assess the Efficacy and Safety of 12 Weeks of Once Daily, Orally Inhaled, Co-administration of Olodaterol 5µg (Delivered by the Respimat® Inhaler) and Tiotropium 18µg (Delivered by the HandiHaler®) Compared to Once Daily, Orally Inhaled, Co-administration of Placebo (Delivered by the Respimat® Inhaler) and Tiotropium 18µg (Delivered by the HandiHaler®) in Patients With Chronic Obstructive Pulmonary Disease (COPD)[ANHELTO TM 1]
Brief Title: Co-administration of Olodaterol Respimat® and Tiotropium Handihaler®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.51
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

ARMS (2):
- Olodaterol and Tiotropium (Experimental): 2 puffs olodaterol from Respimat and one capsule tiotropium from Handihaler once daily in am, co-administered
  Interventions: Drug: Olodaterol; Drug: Tiotropium
- Placebo and Tiotropium (Other): 2 puffs placebo inhalation solution from Respimat and one capsule tiotropium from Handihaler once daily in am, co-administered
  Interventions: Drug: Tiotropium; Drug: Placebo matching Olodaterol

INTERVENTIONS:
Drug: Tiotropium — Marketed dose
  Arms: Placebo and Tiotropium
Drug: Placebo matching Olodaterol — One dose
  Arms: Placebo and Tiotropium
Drug: Olodaterol — One dose
  Arms: Olodaterol and Tiotropium
Drug: Tiotropium — Marketed dose
  Arms: Olodaterol and Tiotropium

SUMMARY:
The overall objective of this study is to assess efficacy and safety of 12 weeks, once daily, orally inhaled co-administration of olodaterol 5 µg (delivered by the Respimat® Inhaler) and tiotropium (delivered by the Handihaler® as Spiriva Handihaler®), compared to tiotropium (Spiriva Handihaler®) monotherapy on lung function in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization-Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions.
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria: Patients must have a relatively stable airway obstruction with a post-bronchodilator FEV1 = 30 % and < 80% of predicted normal and a post-bronchodilator FEV1/FVC <70% at Visit 1.
3. Male or female patients, 40 years of age or older.
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years
5. Patients must be able to: perform technically acceptable pulmonary function tests, and maintain records(paper diary).
6. Patients must be able to inhale medication in a competent manner from the Respimat Inhaler as well as the Handihaler.

Exclusion criteria:

1. Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patients ability to participate in the study.
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an AST >x2 ULN, ALT >x2 ULN, bilirubin >x2 ULN or creatinine >x2 ULN will be excluded regardless of clinical condition (a repeat laboratory evaluation will not be conducted in these patients).
3. Patients with a history of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma. If a patient has a total blood eosinophil count =600/mm3, source documentation is required to verify that the increased eosinophil count is related to a non-asthmatic condition.
4. A diagnosis of thyrotoxicosis (due to the known class side effect profile of ß2-agonists).
5. A diagnosis of paroxysmal tachycardia (>100 beats per minute) (due to the known class side effect profile of ß2-agonists).
6. A history of myocardial infarction within 1 year of screening visit (Visit 1).
7. Unstable or life-threatening cardiac arrhythmia.
8. Hospitalization for heart failure within the past year.
9. Known active tuberculosis.
10. A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed).
11. A history of life-threatening pulmonary obstruction.
12. A history of cystic fibrosis.
13. Clinically evident bronchiectasis.
14. A history of significant alcohol or drug abuse.
15. Patients who have undergone thoracotomy with pulmonary resection (patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1).
16. Patients being treated with oral or patch ß-adrenergics.
17. Patients being treated with oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
18. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigators opinion will be unable to abstain from the use of oxygen therapy during clinic visits.
19. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program.
20. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to screening visit (Visit 1).
21. Patients with known hypersensitivity to ß-adrenergic drugs, BAC, EDTA, or any other component of the Respimat® inhalation solution.
22. Patients with known hypersensitivity to anticholinergic drugs, lactose, or any other components of the HandiHaler®.
23. Pregnant or nursing women.
24. Women of childbearing potential not using a highly effective method of birth control*. Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.

    * as per ICH M3(R2) a highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year).
25. Patients who have previously been randomised in this study or are currently participating in another study.
26. Patients who are unable to comply with pulmonary medication restrictions prior to randomisation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1134 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (90):
- United States (90):
  - 1222.51.01055 Boehringer Ingelheim Investigational Site, Florence, Alabama
  - 1222.51.01087 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1222.51.01066 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1222.51.01069 Boehringer Ingelheim Investigational Site, Scottsdale, Arizona
  - 1222.51.01040 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 1222.51.01064 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 1222.51.01060 Boehringer Ingelheim Investigational Site, Fullerton, California
  - 1222.51.01084 Boehringer Ingelheim Investigational Site, Lincoln, California
  - 1222.51.01041 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1222.51.01094 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1222.51.01015 Boehringer Ingelheim Investigational Site, Torrance, California
  - 1222.51.01052 Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - 1222.51.01010 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1222.51.01042 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1222.51.01070 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1222.51.01006 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1222.51.01021 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1222.51.01082 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1222.51.01065 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1222.51.01051 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1222.51.01092 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1222.51.01081 Boehringer Ingelheim Investigational Site, Ormond Beach, Florida
  - 1222.51.01054 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 1222.51.01062 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1222.51.01088 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1222.51.01079 Boehringer Ingelheim Investigational Site, Tamarac, Florida
  - 1222.51.01075 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1222.51.01076 Boehringer Ingelheim Investigational Site, Austell, Georgia
  - 1222.51.01057 Boehringer Ingelheim Investigational Site, Duluth, Georgia
  - 1222.51.01086 Boehringer Ingelheim Investigational Site, Lawrenceville, Georgia
  - 1222.51.01019 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1222.51.01027 Boehringer Ingelheim Investigational Site, Eagle, Idaho
  - 1222.51.01048 Boehringer Ingelheim Investigational Site, Arlingron Heights, Illinois
  - 1222.51.01044 Boehringer Ingelheim Investigational Site, River Forest, Illinois
  - 1222.51.01043 Boehringer Ingelheim Investigational Site, Skokie, Illinois
  - 1222.51.01090 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1222.51.01023 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1222.51.01071 Boehringer Ingelheim Investigational Site, Opelousas, Louisiana
  - 1222.51.01050 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1222.51.01049 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1222.51.01025 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 1222.51.01078 Boehringer Ingelheim Investigational Site, Edina, Minnesota
  - 1222.51.01033 Boehringer Ingelheim Investigational Site, Fridley, Minnesota
  - 1222.51.01074 Boehringer Ingelheim Investigational Site, Saint Charles, Missouri
  - 1222.51.01037 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1222.51.01039 Boehringer Ingelheim Investigational Site, Reno, Nevada
  - 1222.51.01045 Boehringer Ingelheim Investigational Site, Larchmont, New York
  - 1222.51.01018 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1222.51.01014 Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - 1222.51.01077 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1222.51.01056 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 1222.51.01032 Boehringer Ingelheim Investigational Site, Canton, Ohio
  - 1222.51.01011 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1222.51.01005 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1222.51.01093 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1222.51.01089 Boehringer Ingelheim Investigational Site, Sylvania, Ohio
  - 1222.51.01080 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1222.51.01017 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1222.51.01047 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1222.51.01031 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 1222.51.01020 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1222.51.01053 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1222.51.01016 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 1222.51.01004 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1222.51.01030 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1222.51.01009 Boehringer Ingelheim Investigational Site, Johnston, Rhode Island
  - 1222.51.01036 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1222.51.01061 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1222.51.01038 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1222.51.01046 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 1222.51.01022 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 1222.51.01063 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1222.51.01013 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1222.51.01024 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1222.51.01012 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1222.51.01008 Boehringer Ingelheim Investigational Site, Rapid City, South Dakota
  - 1222.51.01035 Boehringer Ingelheim Investigational Site, Johnson City, Tennessee
  - 1222.51.01028 Boehringer Ingelheim Investigational Site, Boerne, Texas
  - 1222.51.01083 Boehringer Ingelheim Investigational Site, Corsicana, Texas
  - 1222.51.01085 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1222.51.01073 Boehringer Ingelheim Investigational Site, Longview, Texas
  - 1222.51.01003 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1222.51.01058 Boehringer Ingelheim Investigational Site, Murray, Utah
  - 1222.51.01068 Boehringer Ingelheim Investigational Site, Abingdon, Virginia
  - 1222.51.01029 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1222.51.01034 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1222.51.01072 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1222.51.01091 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1222.51.01002 Boehringer Ingelheim Investigational Site, Vancouver, Washington
  - 1222.51.01001 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia

REFERENCES:
- [Derived] ZuWallack R, Allen L, Hernandez G, Ting N, Abrahams R. Efficacy and safety of combining olodaterol Respimat((R)) and tiotropium HandiHaler((R)) in patients with COPD: results of two randomized, double-blind, active-controlled studies. Int J Chron Obstruct Pulmon Dis. 2014 Oct 14;9:1133-44. doi: 10.2147/COPD.S72482. eCollection 2014. PMID 25342898

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1134 patients were entered and randomized to treatment and 1132 patients were treated with study medication.
Groups:
- Olodaterol (5µg) and Tiotropium (18µg): 2 puffs olodaterol from Respimat and one capsule tiotropium from Handihaler once daily in am, co-administered
  Olodaterol: One dose
  Tiotropium: Marketed dose
- Placebo and Tiotropium (18µg): 2 puffs placebo inhalation solution from Respimat and one capsule tiotropium from Handihaler once daily in am, co-administered
  Tiotropium: Marketed dose, 2 inhalations from 1 capsule once daily in the morning
  Placebo matching Olodaterol: One dose, 2 inhalations once daily in the morning
Period: Overall Study
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Started | 567 | 565
Completed | 527 | 525
Not Completed | 40 | 40
Not completed — Adverse Event | 18 | 16
Not completed — Lack of Efficacy | 1 | 0
Not completed — Non compliance protocol | 7 | 6
Not completed — Lost to Follow-up | 2 | 3
Not completed — Consent withdrawn | 7 | 9
Not completed — Other reasons | 5 | 6

BASELINE CHARACTERISTICS:
Population: Treated set (TS), which includes all randomized patients who receive at least one dose of double-blind study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg) | Total
Number analyzed (Participants) | 567 | 565 | 1132
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.1) | 64.8 (9.1) | 64.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 288 | 280 | 568
  Male | 279 | 285 | 564

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-3h Response at 12 Weeks; Defined as Change From Baseline to Week 12
Description: FEV1 (Forced expiratory volume in 1 second) AUC0-3h (area under the curve) response at 12 weeks; defined as change from baseline to Week 12
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks. FAS included all patients in the treated set who had both baseline and at least one post-baseline measurement at or before 12 weeks for any of the co-primary efficacy variables
Measure: Least Squares Mean (Standard Error); unit: Area Under the Curve (L)
Groups:
- Olodaterol (5µg) and Tiotropium (18µg): 2 puffs olodaterol from Respimat and one capsule tiotropium from Handihaler once daily in am, co-administered
  Olodaterol: One dose, 2 inhalations once daily in the morning
  Tiotropium: Marketed dose, 2 inhalations from 1 capsule once daily in the morning
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 563 | 564
Area Under the Curve (L) | 0.313 (0.010) | 0.196 (0.010)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); Results are from an MMRM model. Fixed effects include treatment, visit, treatment by visit interaction, baseline and baseline by visit interaction. Patient is considered random and an unstructured covariance structure was used. Number of patients contributing to models: Tio+Placebo (564), Tio+Olo 5ug (563); Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measure; Mean Difference (Final Values) = 0.117, 95% CI 2-sided [0.090 to 0.144], Standard Error of Mean 0.014

2. Primary Outcome: Trough FEV1 Response at 12 Weeks; Defined as Change From Baseline to Week 12
Description: Trough FEV1 (Forced expiratory volume in 1 second) response at 12 weeks; defined as change from baseline to Week 12
Time Frame: baseline and 12 weeks
Population: Full Analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 548 | 551
L | 0.195 (0.009) | 0.133 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); Results are from an MMRM model. Fixed effects include treatment, visit, treatment by visit interaction, baseline and baseline by visit interaction. Patient is considered random and an unstructured covariance structure was used. Number of patients contributing to models: Tio+Placebo (551), Tio+Olo 5ug (548); Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measure; Mean Difference (Final Values) = 0.062, 95% CI 2-sided [0.037 to 0.088], Standard Error of Mean 0.013

3. Secondary Outcome: Peak FEV1 Response at 12 Weeks - Defined as Change From Baseline
Description: Peak FEV1 (Forced Expiratory Volume in 1 second) response at 12 Weeks - defined as changes from baseline
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 563 | 564
L | 0.389 (0.010) | 0.270 (0.010)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed model repeated measure; Mean change from baseline = 0.119, 95% CI 2-sided [0.090 to 0.147], Standard Error of Mean 0.014

4. Secondary Outcome: FVC AUC0-3h Response at 12 Weeks - Defined as Change From Baseline
Description: Forced Vital Capacity (FVC) AUC0-3h response at 12 weeks - defined as change from baseline.
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 563 | 564
L | 0.438 (0.017) | 0.292 (0.017)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed model repeated measure; Mean difference from Tio + Placebo = 0.146, 95% CI 2-sided [0.100 to 0.192], Standard Error of Mean 0.024

5. Secondary Outcome: Trough FVC Response at 12 Weeks- Defined as Change From Baseline
Description: Trough Forced Vital Capacity (FVC) response at 12 weeks- defined as change from baseline.
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 548 | 551
L | 0.276 (0.016) | 0.213 (0.016)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0047, Mixed model repeated measure; Mean difference from Tio + Placebo = 0.063, 95% CI 2-sided [0.019 to 0.106], Standard Error of Mean 0.022

6. Secondary Outcome: Peak FVC Response at 12 Weeks - Defined as Change From Baseline
Description: Peak FVC response at 12 weeks - defined as change from baseline.
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 563 | 564
L | 0.586 (0.017) | 0.433 (0.017)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed model repeated measure; Mean difference from Tio + Placebo = 0.153, 95% CI 2-sided [0.106 to 0.201], Standard Error of Mean 0.024

7. Secondary Outcome: Rescue Medication Usage - Percentage of Rescue Free Days
Description: Rescue medication usage - the percentage of rescue free days. The percentage of rescue free days is defined as: number of rescue free days divided by total exposure, multiplied by 100%. The baseline for the number of rescue-free days was defined as the number of rescue-free days observed during the last week of the baseline period (i.e., the 7 days prior to administration of the first dose of randomized treatment).
Time Frame: over 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 557 | 561
percentage of days
  Week 1 | 52.633 (1.507) | 48.606 (1.502)
  Week 2 | 54.915 (1.534) | 50.774 (1.528)
  Week 3 | 56.562 (1.565) | 50.262 (1.562)
  Week 4 | 60.580 (1.405) | 55.577 (1.399)
  Week 5 | 60.405 (1.581) | 52.614 (1.572)
  Week 6 | 57.782 (1.632) | 50.547 (1.625)
  Week 7 | 58.642 (1.625) | 50.727 (1.614)
  Week 8 | 58.931 (1.648) | 51.618 (1.636)
  Week 9 | 59.350 (1.652) | 51.399 (1.637)
  Week 10 | 59.991 (1.624) | 52.535 (1.615)
  Week 11 | 59.543 (1.651) | 50.584 (1.643)
  Week 12 | 63.353 (1.553) | 54.894 (1.546)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); Week 12: Results are from non-MMRM ANCOVA models by week with LOCF up to each week. Fixed effects include treatment and baseline. Number of patients contributing to models: Tio+Placebo (561), Tio+Olo 5ug (557); Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean difference from Tio+Placebo Week 12 = 8.459, 95% CI 2-sided [4.159 to 12.759], Standard Error of Mean 2.192

8. Secondary Outcome: Rescue Medication Usage - Mean Weekly Rescue Usage (Total Daily)
Description: Rescue medication usage - mean weekly rescue usage (total daily). The baseline for the rescue use was the mean of the observations during the last week of the baseline period. Administration of rescue medication could occur at any point during the trial as deemed necessary by the patient or the investigator. Open label albuterol MDI (100 μg per puff) was provided as rescue medication . Daily, between clinic visits, patients recorded the number of puffs of albuterol in a paper diary.
Time Frame: over 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: usage (total daily) number of puffs
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 557 | 561
usage (total daily) number of puffs
  Week 1 | 1.760 (0.074) | 2.028 (0.074)
  Week 2 | 1.747 (0.079) | 2.073 (0.079)
  Week 3 | 1.699 (0.079) | 2.094 (0.078)
  Week 4 | 1.730 (0.080) | 2.057 (0.080)
  Week 5 | 1.609 (0.080) | 2.037 (0.079)
  Week 6 | 1.682 (0.085) | 2.047 (0.084)
  Week 7 | 1.657 (0.087) | 2.053 (0.086)
  Week 8 | 1.613 (0.085) | 2.042 (0.084)
  Week 9 | 1.622 (0.084) | 2.056 (0.083)
  Week 10 | 1.571 (0.084) | 2.050 (0.083)
  Week 11 | 1.533 (0.080) | 2.020 (0.079)
  Week 12 | 1.520 (0.082) | 1.998 (0.082)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA; Mean difference from Tio+Placebo Week 12 = -0.478, 95% CI 2-sided [-0.706 to -0.250], Standard Error of Mean 0.116

9. Secondary Outcome: Rescue Medication Usage - Mean Weekly Rescue Usage (Daytime)
Description: Rescue medication usage - Mean weekly rescue usage during daytime hours. Administration of rescue medication could occur at any point during the trial as deemed necessary by the patient or the investigator. Open label albuterol MDI (100 μg per puff) was provided as rescue medication by BI, and only the albuterol MDI provided by BI was allowed for rescue medication use. Daily, between clinic visits, patients recorded the number of puffs of albuterol in a paper diary.
Time Frame: over 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 557 | 561
percentage of days
  Week 1 | 0.392 (0.025) | 0.409 (0.025)
  Week 2 | 0.415 (0.030) | 0.449 (0.029)
  Week 3 | 0.394 (0.028) | 0.437 (0.028)
  Week 4 | 0.393 (0.029) | 0.416 (0.029)
  Week 5 | 0.383 (0.030) | 0.454 (0.030)
  Week 6 | 0.404 (0.031) | 0.447 (0.030)
  Week 7 | 0.402 (0.033) | 0.455 (0.032)
  Week 8 | 0.385 (0.030) | 0.451 (0.030)
  Week 9 | 0.404 (0.031) | 0.457 (0.031)
  Week 10 | 0.390 (0.031) | 0.448 (0.031)
  Week 11 | 0.360 (0.030) | 0.441 (0.029)
  Week 12 | 0.346 (0.029) | 0.429 (0.029)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); Results are from non-MMRM ANCOVA models by week with LOCF up to each week. Fixed effects include treatment and baseline. Number of patients contributing to models: Tio+Placebo (561), Tio+Olo 5ug (557); Test type: Superiority or Other; p = 0.0442, ANCOVA; Mean difference from Tio+Placebo Week 12 = -0.083, 95% CI 2-sided [-0.164 to -0.002], Standard Error of Mean 0.041

10. Secondary Outcome: Rescue Medication Usage - Mean Weekly Rescue Usage (Nighttime)
Description: Rescue medication usage - Mean weekly rescue usage during nighttime hours. Administration of rescue medication could occur at any point during the trial as deemed necessary by the patient or the investigator. Open label albuterol MDI (100 μg per puff) was provided as rescue medication by BI, and only the albuterol MDI provided by BI was allowed for rescue medication use. Daily, between clinic visits, patients recorded the number of puffs of albuterol in a paper diary.
Time Frame: over 12 weeks
Population: Full analysis set (FAS) with last observation carried forward (LOCF) imputation
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Number analyzed (Participants) | 557 | 561
percentage of days
  Week 1 | 1.370 (0.062) | 1.617 (0.061)
  Week 2 | 1.336 (0.064) | 1.620 (0.064)
  Week 3 | 1.309 (0.065) | 1.654 (0.064)
  Week 4 | 1.340 (0.065) | 1.640 (0.065)
  Week 5 | 1.230 (0.066) | 1.581 (0.065)
  Week 6 | 1.285 (0.070) | 1.596 (0.069)
  Week 7 | 1.265 (0.070) | 1.600 (0.069)
  Week 8 | 1.237 (0.070) | 1.587 (0.069)
  Week 9 | 1.597 (0.069) | 1.225 (0.068)
  Week 10 | 1.186 (0.070) | 1.600 (0.069)
  Week 11 | 1.177 (0.067) | 1.581 (0.067)
  Week 12 | 1.178 (0.070) | 1.571 (0.069)
Statistical Analysis 1: Comparison: Olodaterol (5µg) and Tiotropium (18µg) vs Placebo and Tiotropium (18µg); [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < .0001, ANCOVA; Mean difference from Tio+Placebo Week 12 = -0.393, 95% CI 2-sided [-0.586 to -0.200], Standard Error of Mean 0.098

ADVERSE EVENTS:
Time Frame: Adverse events were to be documented throughout the trial, i.e., starting with informed consent and ending 21 days after last administration of trial medication. the duration of treatment was up to 12 weeks.
Arm/Group | Olodaterol (5µg) and Tiotropium (18µg) | Placebo and Tiotropium (18µg)
Serious Adverse Events (participants affected / at risk) | 40/567 | 26/565
Other Adverse Events (participants affected / at risk) | 60/567 | 52/565
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5µg) and Tiotropium (18µg) (N=567) | Placebo and Tiotropium (18µg) (N=565)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Groin infection (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5µg) and Tiotropium (18µg) (N=567) | Placebo and Tiotropium (18µg) (N=565)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 60 | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.